CLINICAL TRIAL: NCT06587880
Title: A Randomized Controlled Trial on the Effect of Different Types of Mouthwash on the Healing of Extraction Sockets
Brief Title: The Effect of Different Types of Mouthwash on Extraction Sockets' Healing
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Ahmad Abdel-Salam Hamdan, Associate Professor, Periodontology, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 224000195; 284/2023-2024 (Other Grant/Funding Number: University of Jordan)
Record Dates: First submitted 2024-08-31; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Extraction Socket Healing; Quality of Life; Postoperative Complications
Keywords: Clinical trial; Mouthwash; Socket healing; Postoperative complications; Quality of life
MeSH Terms: conditions — Postoperative Complications | interventions — chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: The study coordinator will carry out the randomization as mentioned to have a list for the order in which interventions will be given, the same coordinator will prepare opaque bags, then they will move mouthwashes into new opaque bottles and put them in the bags at the same order in the randomization list, instructions sheets will be provided also for the specific mouthwash in the bag.
  The research assistant will have the bags without knowing what is inside them, they will give them to the surgeon after finishing the extraction procedure according to the assigned numbers of the patients which is determined according to the order of visits, the research assistant will leave the surgery room then the surgeon will open the bag to see the instructions to deliver them verbally to the patient and make sure they understand them fully then putting them back in the bag and giving it to the participant.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Bone Bioactive Liquid (Active Comparator): Bone bioactive liquid (BBL) is a saline solution used as a mouthwash that contains calcium chloride (CaCl2) and magnesium dichloride hexahydrate (MgCl2-6H2O) with a net negative charge.
  Interventions: Drug: Bone Bioactive Liquid
- Chlorhexidine Gluconate (Active Comparator): It is a strong bisbiguanide base, with cationic structure at physiological pH (positively charged), and has a broad-spectrum antibacterial activity that works against Gram-positive and Gram- negative bacteria and certain mycetes.
  Interventions: Drug: Chlorhexidine Gluconate
- Warm Saline Mouth Rinse (Active Comparator): Prescribing WSMR as a prophylactic postoperatively is due to the fact that the heat of the solution results in a therapeutic increase in blood flow to the extraction socket.
  Interventions: Drug: Warm Saline Mouth Rinse
- Hyaluronic Acid mouthwash (Active Comparator): It is a high molecular weight non-sulphated polysaccharide. It is biocompatible, non-immunogenic, biodegradable, viscoelastic that make it a preferable biomaterial for medical and pharmaceutical applications without adverse events.
  Interventions: Drug: Hyaluronic Acid mouthwash

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — Prescribed for 7 days period 2 times a day starting 24 hours post-extraction, the patient is instructed to pour 10 ml of the mouthwash into a measuring cup, rinse for 1 minute at an alternative time to teeth brushing. Do not eat or drink for 30 min after use.
  Arms: Chlorhexidine Gluconate
Drug: Bone Bioactive Liquid — Prescribed for 7 days period 2 times a day starting 24 hours post-extraction.
  Arms: Bone Bioactive Liquid
Drug: Hyaluronic Acid mouthwash — Prescribed for 7 days period 3-4 times a day starting 24 hours post-extraction, the patient is instructed to pour 20 ml of the mouthwash into a measuring cup and rinse for 1 minute, at an alternative time to teeth brushing. Do not eat or drink for 30 mins after use.
  Arms: Hyaluronic Acid mouthwash
Drug: Warm Saline Mouth Rinse — Prescribed for 7 days period 2 times a day starting 24 hours post-extraction.
  Arms: Warm Saline Mouth Rinse

SUMMARY:
The goal of this clinical trial is to assess the effect of four different types of mouthwash on socket healing after surgical extractions in male or female patients aged 18 years and older who have a unilateral impacted mandibular third molar indicated for extraction. The main questions it aims to answer are:

The effect of Bone Bioactive Liquid (BBL) mouthwash, Hyaluronic Acid (HA) mouthwash, the Chlorhexidine digluconate (CHX) mouthwash and Warm Saline Mouth Rinse (WSMR) on socket healing after surgical extractions.

The effect of BBL mouthwash, HA mouthwash, the CHX mouthwash and WSMR on patient related factors and their quality of life.

Recruited Participants will be randomized into four intervention groups:

1. First group will receive BBL mouthwash.
2. The second group will receive CHX mouthwash.
3. The third group will be prescribed HA mouthwash.
4. The fourth group will receive Warm Saline Mouth Rinse.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years and older who have a unilateral impacted mandibular third molar that is indicated for extraction with bone removal and the presence of an adjacent second molar.

Exclusion Criteria:

* Soft tissue impaction that will not need any bone removal.
* Presence of any acute oral infection including active Pericoronitis.
* Patients who have undergone radiotherapy in the head and neck region, chemotherapy or systemic long-term corticosteroid treatment.
* Patients receiving medications known to induce gingival hyperplasia; anticonvulsant (phenytoin), immunosuppressant (cyclosporine A), and various calcium channel blockers (nifedipine, verapamil, diltiazem).
* Patients who have taken systemic antibiotics less than 3 months prior to baseline.
* Presence of uncontrolled diabetes, severe nutritional deficiencies and endocrine disturbances.
* Presence of immune deficiency or any immune disease.
* Intravenous bisphosphonates or Oral bisphosphonate intake for more than 3 years.
* Smokers and alcoholics.
* Pregnant or lactating females.
* Hypersensitivity to one of the ingredients listed in any of the mouthwashes, especially chlorhexidine as reactions to this has been reported in the literature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Extraction socket soft tissue healing | Measured at 3, 7, 14 days, 3 and 6 months postoperatively.
  Using a new socket wound healing scale that is a combination of the gingival healing index of Landry et al. and the wound healing scale used by Cervelli et al. to assess the post-extraction wounds in terms of wound dehiscence, epithelialization, quality of granulation tissue filling the post-extraction socket, and depth between early granulation tissue and wound margin.
  A blunt periodontal probe with millimetric markers will be used for this assessment to score a number between 0 (best) and 4 (worst) for the healing socket.

SECONDARY OUTCOMES:
Extraction socket Bone healing | Radiographs will be taken at baseline and at 6 months after extraction.
  Using panoramic radiographs and following the Longitudinal radiographic assessment (LRA) technique categorized as: A. The empty socket is completely radiolucent, and lamina dura is observed clearly around the socket. B. Socket region is hazy and lamina dura is observed around the socket. C. There is a mixed radiolucent-radiopaque appearance inside the socket and lamina dura has been partially disappeared. D. Mature bone is seen inside the socket and lamina dura has disappeared completely (no difference between the socket and normal bone).
The resulting periodontal defect of the adjacent second molar | Preoperatively and at 3, 7, 14 days, 3 and 6 months postoperatively, we may call the patients for further assessment at 9 and 12 months
  Will be evaluated using a UNC 15 perio probe with three clinical parameters: the first is probing depth (PD) measured in mm at three sites of the second molar tooth: Distal (D), disto-buccal (DB), and disto-lingual (DL).
The resulting periodontal defect of the adjacent second molar | Preoperatively and at 3, 7, 14 days, 3 and 6 months postoperatively, we may call the patients for further assessment at 9 and 12 months
  Will be evaluated using a UNC 15 perio probe with three clinical parameters: the second is gingival recession (GR) measured in mm at three sites of the second molar tooth: Distal (D), disto-buccal (DB), and disto-lingual (DL).
The resulting periodontal defect of the adjacent second molar | Preoperatively and at 3, 7, 14 days, 3 and 6 months postoperatively, we may call the patients for further assessment at 9 and 12 months
  Will be evaluated using a UNC 15 perio probe with three clinical parameters: the third is bleeding on probing (BOP) measured as present or not at three sites of the second molar tooth: Distal (D), disto-buccal (DB), and disto-lingual (DL).
Quality of life of the patients (QOL) after extraction | At 3, 7, 14 days, 3 and 6 months postoperatively.
  Assessed based on a questionnaire that addresses different aspects including social and work isolation, ability to eat and speak, impairment of sleep schedule, their physical appearance related to swelling, bleeding and Paresthesia. Answers to the presented questions are in the form of a four-point scale regarding their experience at the time the participants given the form to fill.
Pain at the extraction side | At 3, 7, 14 days, 3 and 6 months postoperatively.
  Assessed using a 10cm long visual analog scale (VAS) where 0= no pain and 10= maximum amount of pain.
Trismus | Pre-operatively and at 3, 7, 14 days, 3 and 6 months postoperatively.
  By measuring the interincisal distance at the maximum mouth opening pre-operatively and at 3, 7, 14 days, 3 and 6 months postoperatively, then the difference between pre- and postoperative will be taken.
Facial swelling at the extraction side | Preoperatively and at 3, 7, 14 days, 3 and 6 months postoperatively.
  Assessed using a soft tape to measure the distance between the lowest point of the tragus and the soft tissue pogonion, the lowest point of the tragus and the lateral corner of the mouth, the lateral corner of the eye and the angle of the mandible. These measurements will be taken preoperatively and at 3, 7, 14 days, 3 and 6 months postoperatively. Then the difference between the pre-operative and postoperative values will be divided by the value obtained in the preoperative period and multiplied by 100 to have the final percentage for the post-operative day.
Socio-demographic factors and medical history | Once preoperatively.
  Data taken from participants using a form.
Peri-operative factors | During the surgical procedure.
  Operation time (min) categorized as <=20, >20 to 30, >30 to 40, >40.
Peri-operative factors | During the surgical procedure.
  Amount of anesthesia administered.
Peri-operative factors | During the surgical procedure.
  Tooth sectioning (done, not done).
Peri-operative factors | During the surgical procedure.
  The surgeon's perception of difficulty categorized as <=9, >9 to 12, >12 to 16, >16.
Pre-operative factors | Once preoperatively.
  The radiographic anatomical relationship between the tooth roots and mandibular canal as it appears on the radiographic image taken preoperatively, categorized as: No association between root structure and the superior border of the canal, Root structure impinging the superior border of canal, Overlapping root structure and canal.
Pre-operative factors | Once preoperatively.
  Prior symptoms related to the third molar to be extracted categorized as: present, absent.
Pre-operative factors | Once preoperatively.
  Indication for the surgical extraction of the third molar categorized as: prophylactic extraction, pain related to the third molar, orthodontic indication.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Hamdan, Ph.D. in Periodontics, Principal Investigator — Faculty of Dentistry - University of Jordan
Locations (1):
- University of Jordan hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share only IPD used in the results publication
Supporting Information: Study Protocol
Time Frame: Beginning from publication with no end date
Access Criteria: The principal investigator will review requests for IPD sharing according to the predetermined set of criteria. The criteria that must be met in order for data to be shared are: having a study protocol that has been approved by an independent review committee identified for IPD meta-analyses. The study protocol must be submitted through email then when reviewed data requestors will need to sign a data access agreement. The data requestor will be provided with the IPD file that can be accessed by them only by having their email listed as a viewer in the sharing list of a folder stored on the DropBox website, this folder has the data excel sheet file and the study protocol as the supporting material.
URL: https://www.dropbox.com/scl/fo/0ku8sqasy9vk6l0c4bs4v/AKSE0PV_oEL48ImAc0lnjhs?rlkey=7ik6ywbm05uvkq7of7s7c1b73&dl=0

REFERENCES:
- [Background] Osunde OD, Adebola RA, Adeoye JB, Bassey GO. Comparative study of the effect of warm saline mouth rinse on complications after dental extractions. Int J Oral Maxillofac Surg. 2014 May;43(5):649-53. doi: 10.1016/j.ijom.2013.09.016. Epub 2013 Dec 5. PMID 24314857
- [Background] Adekunle AA, Egbunah UP, Erinoso OA, Adeyemo WL. Effectiveness of warm saline mouth bath in preventing alveolar osteitis: A systematic review and meta-analysis. J Craniomaxillofac Surg. 2021 Oct;49(10):980-988. doi: 10.1016/j.jcms.2021.09.001. Epub 2021 Sep 4. PMID 34509363
- [Background] Cho H, Lynham AJ, Hsu E. Postoperative interventions to reduce inflammatory complications after third molar surgery: review of the current evidence. Aust Dent J. 2017 Dec;62(4):412-419. doi: 10.1111/adj.12526. Epub 2017 Jun 14. PMID 28498604
- [Background] Maria de Souza G, Elias GM, Pereira de Andrade PF, Andrade Sales KN, Galvao EL, Moreira Falci SG. The Effectiveness of Hyaluronic Acid in Controlling Pain, Edema, and Trismus After Extraction of Third Molars: Systematic Review and Meta-Analysis. J Oral Maxillofac Surg. 2020 Dec;78(12):2154.e1-2154.e12. doi: 10.1016/j.joms.2020.07.005. Epub 2020 Jul 14. PMID 32771444
- [Background] Canellas JVDS, Fraga SRG, Santoro MF, Netto JNS, Tinoco EMB. Intrasocket interventions to prevent alveolar osteitis after mandibular third molar surgery: A systematic review and network meta-analysis. J Craniomaxillofac Surg. 2020 Sep;48(9):902-913. doi: 10.1016/j.jcms.2020.06.012. Epub 2020 Jul 8. PMID 32718882
- [Background] Afat IM, Akdogan ET, Gonul O. Effects of leukocyte- and platelet-rich fibrin alone and combined with hyaluronic acid on early soft tissue healing after surgical extraction of impacted mandibular third molars: A prospective clinical study. J Craniomaxillofac Surg. 2019 Feb;47(2):280-286. doi: 10.1016/j.jcms.2018.11.023. Epub 2018 Dec 3. PMID 30579747
- [Background] Yilmaz N, Demirtas N, Kazancioglu HO, Bayer S, Acar AH, Mihmanli A. The efficacy of hyaluronic acid in postextraction sockets of impacted third molars: A pilot study. Niger J Clin Pract. 2017 Dec;20(12):1626-1631. doi: 10.4103/1119-3077.224131. PMID 29378998
- [Background] Koray M, Ofluoglu D, Onal EA, Ozgul M, Ersev H, Yaltirik M, Tanyeri H. Efficacy of hyaluronic acid spray on swelling, pain, and trismus after surgical extraction of impacted mandibular third molars. Int J Oral Maxillofac Surg. 2014 Nov;43(11):1399-403. doi: 10.1016/j.ijom.2014.05.003. Epub 2014 Jun 10. PMID 24924267
- [Background] Ibraheem W, Jedaiba WH, Alnami AM, Hussain Baiti LA, Ali Manqari SM, Bhati A, Almarghlani A, Assaggaf M. Efficacy of hyaluronic acid gel and spray in healing of extraction wound: a randomized controlled study. Eur Rev Med Pharmacol Sci. 2022 May;26(10):3444-3449. doi: 10.26355/eurrev_202205_28838. PMID 35647824
- [Background] Kim JJ, Song HY, Ben Amara H, Kyung-Rim K, Koo KT. Hyaluronic Acid Improves Bone Formation in Extraction Sockets With Chronic Pathology: A Pilot Study in Dogs. J Periodontol. 2016 Jul;87(7):790-5. doi: 10.1902/jop.2016.150707. Epub 2016 Mar 18. PMID 26991484
- [Background] Gocmen G, Gonul O, Oktay NS, Yarat A, Goker K. The antioxidant and anti-inflammatory efficiency of hyaluronic acid after third molar extraction. J Craniomaxillofac Surg. 2015 Sep;43(7):1033-7. doi: 10.1016/j.jcms.2015.04.022. Epub 2015 May 6. PMID 26027861
- [Background] Rodrigues SV, Acharya AB, Bhadbhade S, Thakur SL. Hyaluronan-containing mouthwash as an adjunctive plaque-control agent. Oral Health Prev Dent. 2010;8(4):389-94. PMID 21180677
- [Background] Romano CL, De Vecchi E, Bortolin M, Morelli I, Drago L. Hyaluronic Acid and Its Composites as a Local Antimicrobial/Antiadhesive Barrier. J Bone Jt Infect. 2017 Jan 1;2(1):63-72. doi: 10.7150/jbji.17705. eCollection 2017. PMID 28529865
- [Background] Phillips C, White RP Jr, Shugars DA, Zhou X. Risk factors associated with prolonged recovery and delayed healing after third molar surgery. J Oral Maxillofac Surg. 2003 Dec;61(12):1436-48. doi: 10.1016/j.joms.2003.08.003. PMID 14663809
- [Background] Sasaki T, Watanabe C. Stimulation of osteoinduction in bone wound healing by high-molecular hyaluronic acid. Bone. 1995 Jan;16(1):9-15. doi: 10.1016/s8756-3282(94)00001-8. PMID 7742090
- [Background] Gizligoz B, Ince Kuka G, Tunar OL, Ozkan Karaca E, Gursoy H, Kuru B. Plaque Inhibitory Effect of Hyaluronan-Containing Mouthwash in a 4-Day Non-Brushing Model. Oral Health Prev Dent. 2020 Feb 14;18(1):61-70. doi: 10.3290/j.ohpd.a43936. PMID 32051972
- [Background] Varoni E, Tarce M, Lodi G, Carrassi A. Chlorhexidine (CHX) in dentistry: state of the art. Minerva Stomatol. 2012 Sep;61(9):399-419. English, Italian. PMID 22976567
- [Background] Ferres-Amat E, Al Madhoun A, Ferres-Amat E, Al Demour S, Ababneh MA, Ferres-Padro E, Marti C, Carrio N, Barajas M, Atari M. Histologic and Histomorphometric Evaluation of a New Bioactive Liquid BBL on Implant Surface: A Preclinical Study in Foxhound Dogs. Materials (Basel). 2021 Oct 19;14(20):6217. doi: 10.3390/ma14206217. PMID 34683810
- [Background] Ferres-Amat E, Al Madhoun A, Ferres-Amat E, Carrio N, Barajas M, Al-Madhoun AS, Ferres-Padro E, Marti C, Atari M. Comparison of 0.12% Chlorhexidine and a New Bone Bioactive Liquid, BBL, in Mouthwash for Oral Wound Healing: A Randomized, Double Blind Clinical Human Trial. J Pers Med. 2022 Oct 16;12(10):1725. doi: 10.3390/jpm12101725. PMID 36294864
- [Background] Oginni FO, Ugboko VI, Assam E, Ogunbodede EO. Postoperative complaints following impacted mandibular third molar surgery in Ile-Ife, Nigeria. SADJ. 2002 Jul;57(7):264-8. PMID 12271954
- [Background] Yamada SI, Hasegawa T, Yoshimura N, Hakoyama Y, Nitta T, Hirahara N, Miyamoto H, Yoshimura H, Ueda N, Yamamura Y, Okuyama H, Takizawa A, Nakanishi Y, Iwata E, Akita D, Itoh R, Kubo K, Kondo S, Hata H, Koyama Y, Miyamoto Y, Nakahara H, Akashi M, Kirita T, Shibuya Y, Umeda M, Kurita H. Prevalence of and risk factors for postoperative complications after lower third molar extraction: A multicenter prospective observational study in Japan. Medicine (Baltimore). 2022 Aug 12;101(32):e29989. doi: 10.1097/MD.0000000000029989. PMID 35960058
- [Background] Araujo MG, Silva CO, Misawa M, Sukekava F. Alveolar socket healing: what can we learn? Periodontol 2000. 2015 Jun;68(1):122-34. doi: 10.1111/prd.12082. PMID 25867983